CLINICAL TRIAL: NCT03763461
Title: Comparison of Pre-warmed, Humidified High Flow Nasal Cannula (HFNC) Oxygen Therapy and Traditional Oxygen Therapy on Patient Comfort and Gas Exchange During Awake Craniotomy - A Single Centre, Prospective, Randomized, Pilot Trial
Brief Title: HFNC During Awake Craniotomy - Impact on Patient Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112229
Record Dates: First submitted 2018-11-26; First posted 2018-12-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Atelectasis; Patient Comfort
Keywords: Awake Craniotomy; HFNC; Oxygen Therapy; Atelectasis; Ultrasound; Patient Comfort
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNC (Experimental): HFNC will be started at flow of 40 L/min and FiO2 of 40%.
  Interventions: Device: HFNC
- Oxygen Mask (Other): Standard non-humidified oxygen therapy via an oxygen mask at 6 l/min will be performed.
  Interventions: Device: Oxygen Mask

INTERVENTIONS:
Device: HFNC — High flow nasal humidified oxygen HFNC is an air-oxygen blender, which provides high flow (up to 60 L/min) of warmed (36°C) and humidified gas through nasal cannula, allowing tighter control of FiO2 from 0.2 to 1.0.
  Arms: HFNC
Device: Oxygen Mask — Application of oxygen during conscious sedation
  Arms: Oxygen Mask

SUMMARY:
Background: Patients undergoing awake brain surgery are exposed to non-humidified, non-warmed oxygen/air mix flow through a face mask for a prolonged duration. This causes increased discomfort, inadequate breathing with the risk for hypoxia perioperatively. Humidified high flow nasal cannula (HFNC) oxygen therapy potentially improves patient comfort, oxygen/air exchange, improves surgical conditions and prevents atelectasis of the lung, compared to traditional oxygen administration using a face mask in patients undergoing awake brain surgery.

Results of this trial will be used to initiate a more extensive, multicenter trial to further characterize the potential impact of HFNC.

DETAILED DESCRIPTION:
Background: Patients undergoing awake brain surgery are exposed to non-humidified, non-warmed oxygen/air mix flow through a face mask for a prolonged duration. This causes increased discomfort, inadequate breathing with the risk for hypoxia perioperatively.

Hypothesis: Humidified high flow nasal cannula (HFNC) oxygen therapy improves patient comfort, oxygen/air exchange, improves surgical conditions and prevents atelectasis of the lung, compared to traditional oxygen administration using a face mask in patients undergoing awake brain surgery.

Methods: After obtaining ethics approval and written informed patient consent, 20 patients undergoing scheduled awake brain surgery will be randomized to either HFNC therapy or standard face mask. Evaluation of patient satisfaction, pain / dry upper airway along with drawing of arterial blood gases to measure oxygen/carbon dioxide content of the blood will be performed during and after the procedure. Lung ultrasound will be performed in the recovery room to determine the presence of atelectasis.

Expected results and Significance: We expect that HFNC improves patient comfort as well as breathing / arterial oxygen content in long-duration awake brain surgery. This could result in higher patient satisfaction, shorter times in PACU, a shorter requirement for oxygen therapy, decreased risk for hypoxia during surgery and better elimination of carbon dioxide - which could lead to better surgical conditions due to softer brain tissue and therefore shorter time for the surgical procedure. Potential positive results of this trial will be used to initiate a more extensive, multicenter trial to further characterize the potential impact of HFNC.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective awake craniotomy

Exclusion Criteria:

* ASA > 4
* pregnant females
* Body Mass Index (BMI) > 40
* elective postoperative mechanical ventilation/conversion to general anesthesia
* denial of consent
* obstructive sleep apnea requiring CPAP
* severe COPD requiring home oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Patient comfort using VAS (1-10) | During surgical procedure, an average of 6 hours
  Patient comfort during awake craniotomy

SECONDARY OUTCOMES:
Gas exchange (blood gas analysis) | During surgical procedure (an average of 6 hours) and 15 minutes after PACU admission
Post-operative pulmonary atelectasis using Ultrasound evaluation | Up to 15 minutes before PACU discharge
Incidence of oxygen desaturation (number of events with SaO2 < 90%) | During surgical procedure, an average of 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No